CLINICAL TRIAL: NCT04519086
Title: The Optimization of a Low-dose Computed Tomography Protocol in Patients With Suspected Uncomplicated Acute Appendicitis and BMI Over 30 kg/m2 (OPTICAP BMI >30)
Brief Title: The Optimization of a Low-dose CT Protocol in Patients With Suspected Uncomplicated Acute Appendicitis and BMI >30
Acronym: OPTICAP>30
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: CT imaging equipment was upgraded during trial enrollment. Old imaging protocols were no longer compatible with new generation CT. As these were not comparable to previous imaging, study was suspended for analysis and reporting of imaging so far.
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Paulina Salminen, MD, PhD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPTICAP BMI >30kg/m2
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Appendicitis; Other and Unspecified Acute Appendicitis; Acute Disease; Gastrointestinal Disease; Intra-abdominal Infection
Keywords: low-dose computed tomography; body mass index; BMI > 30
MeSH Terms: conditions — Appendicitis; Acute Disease; Gastrointestinal Diseases; Intraabdominal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose CT for acute appendicitis in patients with BMI >30 (Experimental): Low-dose computed tomography (CT) vs. standard CT for diagnosing acute uncomplicated appendicitis in patients with BMI > 30 Laparoscopic appendectomy
  Interventions: Radiation: Low-dose CT; Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Radiation: Low-dose CT — Low-dose computed tomography for suspected acute uncomplicated appendicitis in patients with BMI >30
Procedure: Laparoscopic appendectomy — All patients with BMI >30, who are diagnosed with an uncomplicated acute appendicitis on low-dose CT-scan will undergo laparoscopic appendectomy to evaluate the sensitivity and specificity of the CT diagnosis

SUMMARY:
This study focuses on the use of contrast enhanced low-dose CT imaging as a modality to differentiate between uncomplicated and complicated acute appendicitis. Accurate differential diagnosis allows the assessment of all available treatment options. Complicated acute appendicitis requires emergency appendectomy, while uncomplicated acute appendicitis can be safely and efficiently treated with antibiotics in the majority of patients. Our study group already published the results of the initial OPTICAP trial enrolling patients with BMI under 30 showing similar accuracy between the low-dose and the stadard dose CT, but a significant dose reduction associated with the low-dose CT. All patients will undergo both imaging protocols as the standard CT is also optimized for a low as possible radiation dosage and imaging sequence per patient is randomized due to the optimization of contrast media injection timing. All patients participating in this study will be treated operatively with a laparoscopic appendectomy to obtain histological confirmation for the diagnosis to evaluate the accuracy of the CT imaging. The aim of this study is to optimize a well-performing low-dose CT imaging protocol to use in the diagnosis of uncomplicated acute appendicitis in patients with body mass index over 30 kg/m2.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common causes of abdominal pain in emergency departments as well as one of the most common indications for emergency abdominal surgery. The clinical diagnosis has been based on patient history, physical examination and laboratory findings as well as the "clinical eye" of the surgeon. Still the diagnosis remains challenging. One of the main problems is that many other disorders can mimic the clinical presentation of appendicitis, thus increasing the role of imaging techniques to aid in diagnostic accuracy. Now preoperative imaging in patients with suspected acute appendicitis is currently widely accepted as the gold standard and CT has been shown to clearly outperform US in terms of diagnostic performance. Currently CT imaging is considered the primary imaging modality in the diagnosis for acute appendicitis as it is appraised for its high sensitivity and specificity. The main disadvantage of CT imaging is exposure to radiation. Thus the favorable diagnostic performance of CT imaging has encouraged optimization of protocols to minimize exposure to radiation through the development of low-dose CT protocols. Initial studies have indicated that contrast enhanced low-dose CT was not inferior to standard-dose contrast enhanced CT with no statistical significance in negative appendectomy rates, appendiceal perforation rates or patients requiring additional imaging.

This study focuses on the use of contrast enhanced low-dose CT imaging as a modality to differentiate between uncomplicated and complicated acute appendicitis in patients with BMI over 30 kg/m2. Accurate differential diagnosis allows the assessment of all available treatment options. Complicated acute appendicitis requires emergency appendectomy, while uncomplicated acute appendicitis can be safely and efficiently treated with antibiotics in the majority of patients. Our study group already published the results of the initial OPTICAP trial enrolling patients with BMI under 30 showing similar accuracy between the low-dose and the stadard dose CT, but a significant dose reduction associated with the low-dose CT. All patients will undergo both imaging protocols as the standard CT is also optimized for a low as possible radiation dosage and imaging sequence per patient is randomized due to the optimization of contrast media injection timing. All patients participating in this study will be treated operatively with a laparoscopic appendectomy to obtain histological confirmation for the diagnosis to evaluate the accuracy of the CT imaging. The aim of this study is to optimize a well-performing low-dose CT imaging protocol to use in the diagnosis of uncomplicated acute appendicitis in patients with body mass index over 30 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Clinical suspicion of acute uncomplicated appendicitis based on history, physical examination, laboratory findings evaluated by a senior surgeon
* Body mass index over 30 kg/m2

Exclusion Criteria:

* Age <18 years or > 60 years
* Pregnancy or breastfeeding
* Allergy to contrast material or iodine
* History of appendectomy
* Renal failure, creatinine-value greater than the upper reference value
* Diabetes mellitus and metformin medication
* Suspicion of peritonitis and appendiceal perforation
* Incapability to cooperate and give consent to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2023-11-17 (Estimated)

PRIMARY OUTCOMES:
The accuracy of low-dose vs. standard CT in diagnosing acute uncomplicated appendicitis in patients with BMI >30 | 30 days
  CT accuracy between low-dose and standard CT will be evaluated based on the operative and histopathological findings after laparoscopic appendectomy

SECONDARY OUTCOMES:
Negative appendectomy rate | 30 days
Appendiceal perforation rate | 30 days
Sensitivity and specificity of the imaging protocols | 30 days
Radiation dose | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No
Available from the study PI upon request.